CLINICAL TRIAL: NCT04308096
Title: A Phase 3 Long-term Extension Study of KRN23 in Patients With X-linked Hypophosphatemic Rickets/Osteomalacia and a Post-marketing Study of KRN23 Switched From the Phase 3 Long-term Extension Study
Brief Title: A Study of KRN23 in Adult and Pediatric Patients With X-linked Hypophosphatemic Rickets/Osteomalacia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN23-004
Record Dates: First submitted 2020-02-26; First posted 2020-03-13 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: XLH
MeSH Terms: interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KRN23 (Experimental): Subjects will receive subcutaneous injections of KRN23 every 4 weeks (adult) or 2 weeks (pediatric) from Week 0 through Week 140.
  Interventions: Drug: KRN23

INTERVENTIONS:
Drug: KRN23 — The starting dose of KRN23 will be the dose used for the last administration in the preceding studies. The dose may be modified subsequently in accordance with the criteria for dose and dose adjustment.

SUMMARY:
Before switching to the post-marketing study:

Assess the efficacy and safety of KRN23 administered subcutaneously once every 4 or 2 weeks in adult or children with XLH

After switching to the post-marketing study:

To evaluate the safety and efficacy of KRN23, which was switched from the investigational product to the post-marketing investigational product, at the approved dose and dosing regimen in subjects who continued treatment

ELIGIBILITY:
Inclusion Criteria:

1. Personally submitted voluntary written informed consent to participate in the study; For pediatric patients, personally submitted voluntary written informed consent by a legally authorized representative.

   If appropriate, written or verbal assent to participate in the study should be obtained from patients.
2. Patients meeting any of the followings;

   1. For adult XLH patients, completion the final observation at Week 96 in UX023-CL303 or UX023-CL304
   2. For pediatric patients, completion the final observation at Week 64 in UX023-CL301
3. For female patients; women of childbearing potential (except for females who have not reached menarche, permanently sterilized, postmenopausal [12 months with no menses without an alternative medical cause] or anatomically not of childbearing potential) with negative pregnancy test at pre-treatment assessment of Week 0
4. For female patient with childbearing potential, or male patients with reproductive capacity; willingness to use acceptable methods of contraception while participating in the study
5. Willingness and ability to cooperatively complete all study procedures, adhere to the visit schedule and follow the investigator's instructions, as considered by investigator or subinvestigator

Exclusion Criteria:

1. Use of oral phosphate for treating XLH, pharmacologic vitamin D metabolites or analogs, aluminum hydroxide antacids, systemic corticosteroids, acetazolamide, and thiazides within 7 days prior to scheduled initial administration of investigational drug
2. Planned or recommended orthopedic surgery (implantation or removal), including staples, 8 plates or osteotomy, during the study period
3. Blood or blood product transfusion within 60 days prior to scheduled initial administration of investigational drug
4. Use of growth hormone therapy within 12 months prior to scheduled initial administration of investigational drug
5. Use of medication to suppress the secretion of parathyroid hormone (e.g., cinacalcet) within 60 days prior to scheduled initial administration of investigational drug
6. Use of any investigational product (except for investigational product of the preceding study) or investigational medical device within 4 months prior to scheduled initial administration of investigational drug, or requirement for any investigational agent prior to completion of all scheduled study assessments
7. Use of a therapeutic monoclonal antibody other than KRN23 within 90 days prior to scheduled initial administration of investigational drug
8. History of being positive for HIV antibody, HBs antigen and/or HCV antibody
9. Anyone otherwise considered unsuitable for the study by the investigator or subinvestigator

At the time of switching to the post-marketing clinical study:

Subjects eligible for enrollment in the post-marketing clinical study must have met both of the following criteria:

1. Personally submitted voluntary written informed consent to participate in the postmarketing clinical study. For pediatric patients, personally submitted voluntary written informed consent by a legally authorized representative. If appropriate, written or verbal assent to participate in the post-marketing clinical study was to be obtained from subjects.
2. Switching to the post-marketing clinical study was necessary and appropriate for the subject from the viewpoint of efficacy and safety, as judged by the investigator or subinvestigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects for each adverse events | up to week 140
Effect to Body temperature | up to week 140
Effect to Pulse rate | up to week 140
Effect to Respiratory rate | up to week 140
Effect to Systolic blood pressure in sitting position | up to week 140
Effect to Diastolic blood pressure in sitting position | up to week 140
Effect to 12-lead electrocardiogram (ECG) | up to week 140
  The presence of abnormality in the electrocardiogram
Effect to renal ultrasound | up to week 140
  The evaluation to nephrocalcinosis in five grades by renal ultrasound
Effect to Echocardiogram | up to week 140
  The presence of ectopic calcification in the heart by Echocardiogram

SECONDARY OUTCOMES:
Concentration of serum phosphorus | up to week 140
Concentration of serum 1,25(OH)2D | up to week 140
Concentration of urinary phosphorus | up to week 140
Concentration of tubular resorption of phosphorus（TRP） | up to week 140
Concentration of maximum tubular reabsorption of phosphate/glomerular filtration rate (TmP/GFR) | up to week 140
concentration of Carboxy terminal cross-linked telopeptide of type 1 collagen (CTx) (Adult patients with XLH) | up to week 140
concentration of Procollagen type 1 N-propeptide (P1NP) (Adult patients with XLH) | up to week 140
concentration of Bone-specific alkaline phosphatase (BALP)(Adult patients with XLH) | up to week 140
Concentration of serum alkaline phosphatase (ALP) (Pediatric patients with XLH) | up to week 140
Motor functions (6 minutes walk test (6MWT)) | up to week 140
Radiographic findings of fracture and enthesopathy (Adult patients with XLH) | up to week 140
  The presence of radiographic fracture and enthesopathy assessed by X-ray (Adult patients with XLH)
Rickets Severity Score (RSS) (Pediatric patients with XLH) | up to week 140
Radiographic Global Impression of Change (RGI-C)(Pediatric patients with XLH) | up to week 140
Z score of height (LMS method) (Pediatric patients with XLH) | up to week 140

OTHER OUTCOMES:
Pharmacokinetics (Serum KRN23 concentration) | up to week 140
Immunogenicity (Anti-KRN23 Antibody) | up to week 140

CONTACTS AND LOCATIONS:
Locations (10):
- Japan (8):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanagawa Prefectural Hospital Organization Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - National University Corporation Osaka University, Suita, Osaka
  - The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - Toranomon Hospital, Minato-Ku, Tokyo
  - Okayama Saiseikai General Hospital, Okayama
  - Japan Community Health Care Organization Osaka Hospital, Osaka
  - Osaka City University Hospital, Osaka
- South Korea (2):
  - Asan Medical Center, Seoul, Korea
  - Seoul National University hospital, Seoul, Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kubota T, Namba N, Tanaka H, Muroya K, Imanishi Y, Takeuchi Y, Kanematsu M, Sun W, Seino Y, Ozono K. Self-Administration of Burosumab in Children and Adults with X-Linked Hypophosphataemia in Two Open-Label, Single-Arm Clinical Studies. Adv Ther. 2023 Apr;40(4):1530-1545. doi: 10.1007/s12325-022-02412-x. Epub 2023 Jan 31. PMID 36719566